CLINICAL TRIAL: NCT02606760
Title: A Randomized, Double-blind, Vehicle-controlled, Parallel Group Trial to Assess the Efficacy, Safety and Tolerability of P-3073 for Topical Treatment of Nail Psoriasis
Brief Title: Study to Evaluate the Efficacy and Safety of P-3073 Nail Solution in the Treatment of Nails Affected by Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Polichem S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PM1434; 2015-002365-34 (EudraCT Number)
Record Dates: First submitted 2015-11-11; First posted 2015-11-17 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Nail Psoriasis
Keywords: Nail psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- P-3073 (Experimental): P-3073
  Interventions: Drug: P-3073
- vehicle of P-3073 (Placebo Comparator): vehicle of P-3073
  Interventions: Drug: Vehicle of P-3073

INTERVENTIONS:
Drug: P-3073
  Arms: P-3073
Drug: Vehicle of P-3073
  Arms: vehicle of P-3073

SUMMARY:
The purpose of this study is to confirm the clinical efficacy and the safety of P-3073 in patients affected by isolated psoriatic nail(s) and/or those with psoriatic nails and concomitant mild to moderate plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent before starting any study related procedures
* Patients aged 18 to 80 years old of any race.
* Males or females.
* Patients with mild to moderate psoriastic fingernail(s) defined as fingernail/s with matrix psoriasis NAPSI score and/or bed psoriasis NAPSI score ≥ 1 and ≤ 3 at baseline.
* In case of skin involvement, patients with established clinical diagnosis of mild-to-moderate psoriasis (BSA involvement ≤ 8% or PASI ≤ 10)

Exclusion Criteria:

* Woman who is pregnant, nursing an infant, or planning a pregnancy during the study period.
* Use of any systemic treatment for psoriasis during the last six months before the screening visit.
* Use of photochemotherapy or other forms of radiotherapy during the last four weeks before the screening visit.
* Positive mycology findings
* Systemic use of immunosuppressives, chemotherapy and corticosteroids during last three months before the screening visit.
* Consumption of Vitamin D or its analogues during the last three months.
* History of hypercalcaemia or hypercalciuria.
* HIV infection or any other immunodeficiency.
* Alcohol or substance abuse.
* Patients with history of allergic reactions to calcipotriol or its excipients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Change in total Nail Psoriasis Severity Index (NAPSI) | Baseline - Week 24

SECONDARY OUTCOMES:
Change in NAPSI matrix | Baseline - Week 24
Change in NAPSI bed | Week 24
Nail Physician Global Assessment (PGA) response rate | Week 24
Change in patient's quality-of-life by means of the Dermatology Life Quality Index (DLQI) | Baseline - Week 24
Change in discomfort by means of the Visual Analogue Scale (VAS) | Week 24
Proportions of nails with improvement in total NAPSI | Week 24
Proportions of nails with improvement in NAPSI Matrix | Week 24
Proportions of nails with improvement in NAPSI bed | Week 24
Overall safety by recording any AE during the entire study duration and the local tolerability by means of severity scores for skin irritation. | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Caserini, MD, Study Director — Polichem S.A.
Locations (7):
- Multiple Locations, Bulgaria
- Multiple Locations, Czechia
- Multiple Locations, Germany
- Multiple Locations, Greece
- Multiple Locations, Latvia
- Multiple Locations, Poland
- Multiple Locations, Russia